CLINICAL TRIAL: NCT02242526
Title: Biologic Versus Synthetic Mesh for Treatment of Paraesophageal Hernia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SB-568818
Record Dates: First submitted 2014-09-03; First posted 2014-09-17 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hiatal Hernia
Keywords: hiatal hernia, recurrence, biologic mesh, synthetic mesh
MeSH Terms: conditions — Hernia, Hiatal; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parietex™ Composite Hiatal Mesh, North Haven, CT (Active Comparator): Synthetic prosthetic mesh Parietex™ Composite Hiatal (PCO 2H) Mesh (Covidien, North Haven, CT) designed for hiatal hernia repair.
  Interventions: Device: Parietex™ Composite Hiatal Mesh, North Haven, CT; Device: Biodesign™ Surgisis® Graft, Cook Medical, Bloomington
- Biodesign™ Surgisis® Graft, Cook Medical, Bloomington (Active Comparator): Biologic mesh Biodesign™ Surgisis® Graft Reinforcement in Hiatal, Cook Medical, Bloomington, IN which will be placed for repair of hiatal hernia
  Interventions: Device: Parietex™ Composite Hiatal Mesh, North Haven, CT; Device: Biodesign™ Surgisis® Graft, Cook Medical, Bloomington

INTERVENTIONS:
Device: Parietex™ Composite Hiatal Mesh, North Haven, CT — Parietex™ Composite Hiatal Mesh (North Haven, CT) designed for hiatal hernia repair.
Device: Biodesign™ Surgisis® Graft, Cook Medical, Bloomington — Biodesign™ Surgisis® Graft (Cook Medical, Bloomington) designed for hiatal hernia repair.

SUMMARY:
The investigators propose a randomized, single blinded controlled trial to compare the use of synthetic versus biologic mesh in hiatal hernia repair, two currently accepted standard of care surgical modalities. The investigators hypothesize that use of synthetic mesh will have lower recurrence at these time points compared to use of biologic mesh.

DETAILED DESCRIPTION:
Patients will be randomized to either a synthetic (light weight synthetic or biologic (small intestinal submucosa ) mesh group. Endpoints will be measured up to 5 years for the study as a whole, at 6 months and at 60 months. Prior to and following laparoscopic paraesophageal hernia repair, patients will be followed with both subjective and objective measures. Subjective evaluation will include symptomatic/quality of life assessment at 1-, 6-, 24-, and 60- month periods; objective evaluation will include Upper GI study /pH probe study for symptomatic patients and for all patients at 6 and 60 months. The investigators hypothesize that use of synthetic mesh will have lower recurrence at these time points compared to use of biologic mesh.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* Age>18 years
* Absence of chronic medical conditions that will affect the quality of life survey, such as fibromyalgia, SLE, Crohn's disease, etc.
* Able to give informed consent
* Able and willing to participate in follow-up evaluations
* Upper GI with a documented hiatal hernia greater than 5cm
* Paraesophageal hernia with clinically relevant symptoms such as heartburn, chest pain, regurgitation, dysphagia, postprandial abdominal pain, shortness of breath, or early satiety.

Exclusion Criteria:

* Previous surgery of the esophagus and/or the stomach
* Emergent operation for acute gastric volvulus or strangulation
* Biopsy consistent with malignancy
* Body Mass Index (BMI) over 35kg/m2
* Inability to perform primary closure of crura
* Active smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Assess for reappearance of hiatal hernia and reflux | 6 months, 60 months
  Change at 6 and 60 months will be assessed by pH and Upper GI (endoscopy) studies to assess for reappearance of hiatal hernia and reflux.

SECONDARY OUTCOMES:
Quality of Life questionnaire | Quality of Life will be assessed at these time periods after the hernia repair 1, 6, 24, and 60 months
  Quality of life questionnaire containing 36 questions

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States